CLINICAL TRIAL: NCT00431106
Title: A Multicenter Randomized Phase III Study of Combination Treatment With Vinorelbine and Gemcitabine Versus Capecitabine Monotherapy in Metastatic Breast Cancer Patients Following Treatment Failure With the Combination of a Taxane and an Anthracycline
Brief Title: Vinorelbine and Gemcitabine Versus Capecitabine in Pretreated Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: D. Mavrudis, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/02.11
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Chemotherapy; Vinorelbine; Gemcitabine; Capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Capecitabine; Vinorelbine

ARMS (2):
- 1 (Active Comparator): Vinorelbine/Gemcitabine (VG)
  Interventions: Drug: Gemcitabine; Drug: Vinorelbine
- 2 (Active Comparator): Capecitabine (Cap)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine at the dose of 1000 mg/m2 intravenously (IV) every 2 weeks for 12 consecutive cycles
  Other Names: Gemzar
  Arms: 1
Drug: Capecitabine — Capecitabine at the dose of 1250 mg/m2 twice daily orally (os), from day 1 to day 14, every 3 weeks for 6 consecutive cycles
  Other Names: Xeloda
  Arms: 2
Drug: Vinorelbine — Vinorelbine at the dose of 25 mg/m2 IV on day 1 every 2 weeks for 12 consecutive cycles
  Other Names: Navelbine
  Arms: 1

SUMMARY:
The combination of vinorelbine and gemcitabine seems to be an important part of the chemotherapy regimens used in metastatic breast cancer patients following treatment failure with the combination of a taxane and an anthracycline. Capecitabine rescue monotherapy in metastatic breast cancer patients following treatment failure with the combination of a taxane and an anthracycline, also seems to be an important part of the chemotherapy regimens used in metastatic breast cancer patients. Whether the combination of vinorelbine and gemcitabine or capecitabine administration is preferable is not yet known, especially in patients with metastatic disease.

DETAILED DESCRIPTION:
This trial will compare the efficacy of combination treatment with Vinorelbine and Gemcitabine versus Capecitabine monotherapy in metastatic breast cancer patients following treatment failure with the combination of a taxane and an anthracycline.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-75 years.
* Performance status World Health Organization (WHO) 0-2.
* Histologically confirmed breast adenocarcinoma.
* Clinical or radiological evidence of metastatic disease that has progressed after combination treatment of a taxane and an anthracycline (Taxotere + Mitoxantrone or Taxotere + Farmorubicine).
* Measurable disease.
* No metastatic central nervous system (CNS) disease.
* Less than 25% of myeloproductive bone marrow irradiated.
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9 gr/mm^3).
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2 mg/dl).
* Informed consent.

Exclusion Criteria:

* Pregnancy or nursing.
* Positive pregnancy test.
* Psychiatric illness or social situation that would preclude study compliance.
* Other concurrent uncontrolled illness.
* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer.

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2002-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression between the two treatment arms | 1 year

SECONDARY OUTCOMES:
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dept. of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dept. of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dept. of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dept. of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dept. of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dept. of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dept. of Medical Oncology, Thessaloniki